CLINICAL TRIAL: NCT03752541
Title: Efficacy and Safety Evaluation of BCMA-UCART（Allogeneic Engineered T-cells Expressing Anti-BCMA Chimeric Antigen Receptor）in the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: Efficacy and Safety Evaluation of BCMA-UCART
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: decided by the sponsor
Sponsor: Bioray Laboratories (Industry)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-CAR-00CH3
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: 0.5-1*10~6/KgBW, 1-2*10~6/KgBW,2-3*10~6/KgBW
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA-UCART (Experimental): Each subject will accept one of the following dosages of BCMA-UCART cells intravenously (IV) on day 0: 0.5-1*10~6/KgBW, 1-2*10~6/KgBW,2-3*10~6/KgBW.
  Interventions: Biological: BCMA-UCART

INTERVENTIONS:
Biological: BCMA-UCART — A conditioning therapy with cyclophosphamide and fludarabine will be conducted for subjects before CART therapy.

SUMMARY:
This trial aims to evaluate the safety and efficacy of BCMA-UCART in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
BCMA(B-Cell maturation antigen) is a tumor antigen of multiple myeloma. Using a genetic engineering strategy to assemble an anti-BCMA CAR(chimeric antigen receptor) in T cells will help these CART cells to recognize and kill BCMA-expressing MM tumor cells. BCMA-UCART is a kind of allogeneic CART, originating from T cells of health donors. This open-label, dose-escalation study aims to evaluate the safety and anti-tumor efficacy of BCMA-UCART in treating relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Have the capacity to give informed consent;
* Confirmed diagnosis of active MM as defined by NCCN and IMWG criteria;
* Have a diagnosis of BCMA+ multiple myeloma (MM), (≥ 5% BCMA+ in CD138+ plasma cells by flow cytometry obtained within 45 days of study enrollment);
* Refractory and relapsed MM patients after > 2 cycles of induction therapy,or,have relapsed or treatment refractory disease following autologous stem cell transplant (ASCT);
* ECOG score=0-2.
* Subjects according with any of the following options:

  * Age≥50;
  * Failure with separation of T cells during autologous CART processing; or,
  * Failure with expansion of autologous CART; or,
  * The proportion of T cells in PBMC <10%; or,
  * Won't benefit from autologous CART therapy because of disease progress.

Exclusion Criteria:

* Pregnant or nursing women; Women of reproductive potential must have a negative serum pregnancy test performed within 48 hours of starting conditioning chemotherapy
* Active infection, HIV infection, syphilis serology reaction positive;
* Active hepatitis B, hepatitis C at the time of screening
* Significant hepatic dysfunction as following, SGOT(serum glutamic-oxaloacetic transaminase)> 5 x upper limit of normal; bilirubin > 3.0 mg/dL;
* Lymphotoxic chemotherapeutic agents within 2 weeks of leukapheresis
* serious mental disorder;
* With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* Participate in other clinical research in the past three months; previously treatment with any gene therapy products
* Contraindication to cyclophosphamide or fludarabine chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 90 days after T cell infusion
  Proportion of patients in whom a response among complete response or partial response, as defined by International Myeloma Working group(IMWG) response criteria , will be observed.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events as a Measure of Safety and Tolerability | Up to 35 days after T cell infusion
  Adverse events assessed according to NCI-CTCAE v4.03 criteria
Duration of persistence of BCMA-UCART | Baseline up to 1 year
  Detect the duration of BCMA-UCART after injection using FACS or Q-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Aibin Liang, PhD, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No